CLINICAL TRIAL: NCT00177099
Title: Neurotrophic Effects of Immunophilin Ligands on Human Hair Follicles Grafted Onto Service Combined Immunodeficient (SCID) Mice
Brief Title: Effects of Ligands on Human Hair Follicles Grafted Onto SCID Mice
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hordinsky, Maria K., MD (Individual)
Organization: University of Minnesota (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0306M49486
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2006-11-13 (Estimated); Status verified 2006-11

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia | interventions — Tacrolimus

INTERVENTIONS:
Drug: FK506, GP11046, GP11511

SUMMARY:
The purpose of this study is to determine if immunophilin ligands may have the potential to reverse hair loss.

DETAILED DESCRIPTION:
Preliminary experiments in C57BL/6J mice showed that immunophilin ligand FK506 and its non-immunosuppressive analogs, GP11046 and GP11511 were capable of promoting telogen to anagen transition. Since GP11046 and GP11511 possess the neurotrophic properties of FK506 without its immunosuppressant capability, the neural action of these immunophilin ligands may play an important role in the hair cycle. This finding has significant clinical implications in that immunophilin ligands may have the potential to reverse alopecia. To further investigate this possibility we propose to explore the response of transplanted miniaturized scalp hair follicles to topically applied immunophilin ligands.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men ages 18-65 with Hamilton type IV or V alopecia

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2003-07; Study Completion 2004-09

PRIMARY OUTCOMES:
The average number of terminal hairs per graft will be compared between the control and the treated group.

SECONDARY OUTCOMES:
The number of follicles in anagen, catagen and telogen per graft will be averaged for each group. The results will be compared between the control and the treated groups.

CONTACTS AND LOCATIONS:
Overall Officials: Marna Ericson, Ph D, Principal Investigator — University of Minnesota; Maria Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States